CLINICAL TRIAL: NCT02028403
Title: Safety, Pharmacokinetics and Immunotherapeutic Activity of an Anti-PD-L1 Antibody (BMS-936559) in HIV-1 Infected Participants on Suppressive cART: A Phase I, Double-Blind, Placebo-Controlled, Ascending Single Dose Study
Brief Title: Safety and Immune Response of BMS-936559 in HIV-Infected People Taking Combination Antiretroviral Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A5326; 11921 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2014-01-03; First posted 2014-01-07 (Estimated); Last update posted 2021-11-05 (Actual); Status verified 2016-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — BMS-936559

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Cohort 1A: single dose 0.3 mg/kg BMS-936559 (Experimental): Participants will receive 0.3 mg/kg of BMS-936559, administered as a single infusion once at study entry.
  Interventions: Drug: BMS-936559
- Cohort 1B: single dose placebo for BMS-936559 (Placebo Comparator): Participants will receive placebo for BMS-936559, administered as a single infusion once at study entry.
  Interventions: Drug: Placebo for BMS-936559
- Cohort 2A: single dose 1 mg/kg BMS-936559 (Experimental): Participants will receive 1 mg/kg of BMS-936559, administered as a single infusion once at study entry.
  Interventions: Drug: BMS-936559
- Cohort 2B: single dose placebo for BMS-936559 (Placebo Comparator): Participants will receive placebo for BMS-936559, administered as a single infusion once at study entry.
  Interventions: Drug: Placebo for BMS-936559
- Cohort 3A: single dose 3 mg/kg BMS-936559 (Experimental): Participants will receive 3 mg/kg of BMS-936559, administered as a single infusion once at study entry.
  Interventions: Drug: BMS-936559
- Cohort 3B: single dose placebo for BMS-936559 (Placebo Comparator): Participants will receive placebo for BMS-936559, administered as a single infusion once at study entry.
  Interventions: Drug: Placebo for BMS-936559
- Cohort 4A: single dose 10 mg/kg BMS-936559 (Experimental): Participants will receive 10 mg/kg of BMS-936559, administered as a single infusion once at study entry.
  Interventions: Drug: BMS-936559
- Cohort 4B: single dose placebo for BMS-936559 (Placebo Comparator): Participants will receive placebo for BMS-936559, administered as a single infusion once at study entry.
  Interventions: Drug: Placebo for BMS-936559

INTERVENTIONS:
Drug: BMS-936559 — 0.3 mg/kg, 1 mg/kg, 3 mg/kg, or 10 mg/kg of BMS-936559, depending on which cohort participants are enrolled in, administered as an intravenous (IV) infusion
  Arms: Cohort 1A: single dose 0.3 mg/kg BMS-936559; Cohort 2A: single dose 1 mg/kg BMS-936559; Cohort 3A: single dose 3 mg/kg BMS-936559; Cohort 4A: single dose 10 mg/kg BMS-936559
Drug: Placebo for BMS-936559 — Sodium chloride for injection 0.9%, USP, administered as an IV infusion
  Arms: Cohort 1B: single dose placebo for BMS-936559; Cohort 2B: single dose placebo for BMS-936559; Cohort 3B: single dose placebo for BMS-936559; Cohort 4B: single dose placebo for BMS-936559

SUMMARY:
People infected with HIV may have low levels of the virus in their body, even if they are taking HIV medications. This study will evaluate the safety, pharmacokinetics (PK) (which is how the body interacts with drugs), and immune response to BMS-936559, a drug that will be administered by an intravenous (IV) infusion, in HIV-infected people receiving combination antiretroviral therapy (cART) who have viral load levels below the limit of detection.

DETAILED DESCRIPTION:
People infected with HIV who are taking cART and have low viral load levels may still have reservoirs of HIV remaining in their body. BMS-936559 is a drug that has been studied in previous clinical trials to treat various types of cancer. The purpose of this study is to evaluate the safety, PK, and immunotherapeutic activity of a single dose of BMS-936559 (administered by an IV infusion) in HIV-infected people who are receiving cART and who have viral loads below the limit of detection. Researchers will also evaluate whether BMS-936559 can reduce hidden reservoirs of HIV.

Participants will be enrolled in four cohorts. Within each cohort, participants will be randomly assigned to receive BMS-936559 (Cohort 1: 0.3 mg/kg; Cohort 2: 1 mg/kg; Cohort 3: 3 mg/kg; or Cohort 4: 10 mg/kg) or placebo. The four cohorts will be enrolled sequentially, with researchers reviewing safety data of the cohort before enrolling participants in the next cohort.

Prior to study entry, all participants must have an eye exam and an electrocardiogram (ECG). At study entry, participants will undergo a medical and medication history review, physical examination, an eye exam, and a blood collection. Some female participants will have a pregnancy test. All participants will then receive a single IV infusion of their assigned dose of BMS-936559 or placebo. The infusion will occur over a period of 60 minutes, and participants will remain in the clinic for observation for an additional 12 hours. Additional study visits will occur at Days 3, 7, 14, 28, and Weeks 10, 16, 24, 36, and 48. These study visits may include a physical examination, blood collection, adherence assessments, and PK evaluations. Some participants may have additional eye exams during the study, on an as-needed basis.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA assay. More information on this criterion is available in the protocol.
* Receiving a stable cART regimen containing at least three agents (not including ritonavir if less than a 200 mg total daily dose) with no changes in the components of their antiretroviral therapy for at least 90 days prior to study entry. NOTE: One of the agents must include an integrase inhibitor, a non-nucleoside reverse transcriptase inhibitor (NNRTI), or a boosted protease inhibitor (PI).
* CD4 cell count greater than or equal to 350 cells/mm^3 obtained within 90 days prior to study entry at any U.S. laboratory that has a clinical laboratory improvement amendments (CLIA) certification or its equivalent
* Plasma HIV-1 RNA below detected limit obtained by Food and Drug Administration (FDA)-approved assays (limit of detection: 75, 50, 40, or 20) for greater than or equal to 2 years on cART. Participants must have at least one documented HIV-1 RNA less than the limit of detection 12-24 months prior to screening and one HIV-1 RNA less than the limit of detection within 12 months prior to screening. NOTE: A single unconfirmed plasma HIV-1 RNA greater than the limit of detection but less than 1,000 copies/mL is allowed if followed by HIV-1 RNA below detectable limits, but none in the 6 months prior to screening.
* Plasma HIV-1 RNA level of less than 40 copies/mL obtained by the Abbott m2000 assay or less than 20 copies/mL by the Roche Taqman v2.0 assay within 90 days prior to entry. The protocol team should be notified as soon as possible if the HIV-1 RNA level is above the limit of detection for either assay.
* Plasma HIV-1 RNA greater than or equal to 0.4 copies/mL by single copy assay (SCA) within 120 days prior to entry
* The following laboratory values obtained within 60 days prior to entry by any U.S. laboratory that has a CLIA certification or its equivalent:

  * Absolute neutrophil count (ANC) greater than or equal to 1,000 cells/mm^3
  * Hemoglobin greater than or equal to 14.0 g/dL for men and greater than or equal to 12.0 g/dL for women
  * Platelet count greater than or equal to 75,000/mm^3
  * Creatinine clearance greater than or equal to 50 mL/min estimated by the Cockcroft-Gault equation. NOTE: A program for calculating creatinine clearance by the Cockcroft-Gault method is available on www.fstrf.org.
  * Alanine aminotransferase (ALT) (SGPT) less than or equal to 2.5 times upper limit of normal (ULN)
  * A.M. cortisol within normal limits
  * Fasting blood sugar within normal limits
  * Total bilirubin less than or equal to 1.6 x ULN. NOTE: If the participant is on an atazanavir-containing therapy then a direct bilirubin should be measured instead of the total bilirubin and must be less than or equal to 1.0 mg/dL.
* The following laboratory values obtained within 90 days prior to entry by any U.S. laboratory that has a CLIA certification or its equivalent:

  * Thyroid stimulating hormone (TSH) and free T4 level within normal limits
  * Hemoglobin A1c (HgbA1c) within normal limits
* Hepatitis C virus (HCV) antibody negative result within 90 days prior to study entry or, if the HCV antibody result is positive, a negative HCV RNA result prior to study entry. Participants who have received HCV treatment in the last 5 years will be excluded.
* Negative hepatitis B surface antigen (HBsAg) result obtained within 90 days prior to study entry
* Karnofsky performance score greater than or equal to 90 within 60 days prior to entry
* Documentation of the availability of the stored pre-entry plasma specimens for HIV-1 RNA SCA determination and stored pre-entry peripheral blood mononuclear cell (PBMC) specimens for CD8 T-cell assays. Sites must receive confirmation from the processing lab via phone, e-mail, or fax, that specimens have been entered into the AIDS Clinical Trials Group's (ACTG's) Laboratory Data Management System (LDMS).
* Ability and willingness of participant or legal guardian/representative to provide informed consent
* Ability and willingness of participant to continue cART throughout the study
* Ability to construct a fully active alternative cART regimen in the event of virologic failure on the current ART regimen
* An ophthalmology exam within 180 days prior to entry and a copy of the results of the exam. NOTE: Ophthalmologic exams done to meet enrollment criteria must be performed by a licensed ophthalmologist within 180 days of the study entry visit. Results of the exam must be available for review and made part of the clinical record.

Exclusion Criteria:

* History of malignancy within the last 5 years or current malignancy requiring cytotoxic therapy. NOTE: A history of non-melanoma skin cancer (e.g., basal cell carcinoma or squamous cell skin cancer) is not exclusionary.
* History of HIV-related opportunistic infections within the last 5 years. More information on this criterion is available in the protocol.
* Current chronic, acute, or recurrent bacterial, fungal, or viral (other than HIV) infections that are serious, in the opinion of the site investigator, and required systemic therapy within 30 days prior to entry
* History of or active autoimmune disorders including but not limited to inflammatory bowel diseases, scleroderma, severe psoriasis, myocarditis, uveitis, pneumonitis, systemic lupus erythematosus, rheumatoid arthritis, optic neuritis, myasthenia gravis, adrenal insufficiency, hypothyroidism and/or hyperthyroidism, autoimmune thyroiditis, or sarcoidosis. More information on this criterion is available in the protocol.
* History of inflammatory disorders of the eye including uveitis (iritis, endophthalmitis, scleritis, retinitis - including viral or other infectious retinitis) and chronic or recurrent post-operative inflammation. NOTE: A history of self-limited conjunctivitis, blepharitis, or hordeolum (stye) are NOT exclusions.
* Previous ocular treatment with silicone oil tamponade (for complex retinal detachment)
* Intraocular surgery within 90 days prior to entry or the anticipated need for intraocular surgery during the course of the study
* Intraocular laser or cryotherapy within 90 days prior to entry or the anticipated need for intraocular laser or cryotherapy during the course of the study
* Evidence on eye exam of active or previous ocular inflammation or uveitis
* Previous history of serious ocular trauma (e.g., penetrating trauma of the eye)
* Severe cataract or other ocular abnormality that precludes adequate examination of the posterior chamber and fundus
* Active infection or inflammation of the eye within 30 days prior to entry that requires systemic or topical therapy or, in the opinion of the site investigator, would complicate on-study evaluation and patient safety. NOTE: A history of self-limited allergic conjunctivitis is NOT an exclusion. More information on this criterion is available in the protocol.
* Immune deficiency other than HIV
* Breastfeeding
* Known allergy/sensitivity or any hypersensitivity to components of BMS-936559 (anti-PD-L1) or its formulation
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Acute or serious illness, in the opinion of the site investigator, requiring systemic treatment and/or hospitalization within 30 days prior to entry
* Use of immunomodulators (e.g., interleukins, interferons, cyclosporine), HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy within 60 days prior to study entry. NOTE: Participants receiving stable physiologic glucocorticoid doses, defined as prednisone less than or equal to 10 mg/day or the equivalent, will not be excluded. Stable physiologic glucocorticoid doses should not be discontinued for the duration of the study. In addition, participants receiving inhaled or topical corticosteroids will not be excluded.
* Intent to use immunomodulators (e.g., IL-2, IL-12, interferons, or tumor necrosis factor [TNF] modifiers) during the course of the study
* Any vaccination within 30 days prior to screening SCA, pre-entry, or entry. Individuals who require vaccination will delay screening SCA until 30 days post-vaccination. Alternatively, vaccinations can occur following the screening SCA, provided they occur greater than or equal to 30 days prior to pre-entry or entry.
* Current HCV antiviral therapy or participants who have received HCV treatment in the last 5 years
* Positive tuberculosis (TB) purified protein derivative (PPD) skin test or interferon-gamma release assay (IGRA) at screening. NOTE: Participants with a prior positive PPD or IGRA who have not completed prophylaxis treatment will be excluded.
* Women of reproductive potential. More information on this criterion is available in the protocol.
* History of chronic obstructive pulmonary disease (COPD)
* Type I and type II diabetes mellitus
* Participants weighing less than 50 kg or greater than 200 kg. NOTE: For participants weighing between 50 kg to 52.9 kg, sites must consult with the A5326 protocol team prior to enrollment. The allowable blood volume to be drawn in an 8-week period for these participants may be less than participants weighing greater than or equal to 53 kg.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Occurrence of a Grade 3 or greater adverse event (AE), including sign/symptom, lab toxicity, or clinical event that is definitely, probably, or possibly related to study treatment | Measured through Day 28
  As judged by the core team, blinded to treatment arm; any time from study treatment administration until 28 days after the administration.
Occurrence of a Grade 1 or > AE of all incident adrenal insufficiency or adrenal crisis (confirmed), myocarditis, pneumonitis, uveitis, immune-mediated hyperthyroidism or hypothyroidism, that is definitely, probably, or possibly related to study | Measured through Day 28
  As judged by the core team, blinded to treatment arm; any time from study treatment administration until 28 days after the administration.
  (Pneumonitis is Category A, B, or C)
Frequency of HIV-1 Gag-specific CD8 T-cells by intracellular staining for interferon (IFN)-gamma at baseline and after treatment (through Day 28) | Measured through Day 28
HIV-1 RNA by single copy assay (SCA) at baseline and after treatment (through Day 28) | Measured through Day 28

SECONDARY OUTCOMES:
PK parameters from non-compartmental analysis (area under curve [AUC], Cmax, V, Tmax, CL/F, t1/2) | Measured through Week 48
Exploratory pharmacodynamic parameters (Emax, EC50) | Measured through Week 48
HIV-1 DNA at baseline and after treatment | Measured through Week 48
Programmed cell death 1 ligand 1 (PD-L1) receptor occupancy | Measured through Week 48
Proportion of total and HIV-1 gag-specific CD8 T-cells expressing programmed cell death 1 (PD-1), PD-L1, and other exhaustion markers | Measured through Week 48
CD107a mobilization and carboxyfluorescein diacetate succinimidyl ester (CFSE) dilution of HIV-1 gag-specific CD8 T-cells | Measured through Week 48
Polyfunctionality of HIV-1 specific CD8 and CD4 T-cells | Measured through Week 48
CD38 and human leukocyte antigen-DR (HLA-DR) expression on CD8 T-cells | Measured through Week 48
Gene expression profiles in whole blood | Measured through Week 48
Detection of antibody to study treatment in plasma | Measured through Week 48
Occurrence of a Grade 3 or greater AE, including sign/symptom, lab toxicity, or clinical event that is definitely, probably, or possibly related to study treatment | Measured through Week 48
  As judged by the core team, blinded to treatment arm; any time greater than or equal to 29 days after the study treatment administration
Occurrence of a Grade 1 or > AE of all incident adrenal insufficiency or adrenal crisis (confirmed), myocarditis, pneumonitis, uveitis, immune mediated hyperthyroidism or hypothyroidism, that is definitely, probably, or possibly related to study | Measured through Week 48
  As judged by the core team, blinded to treatment arm; any time greater than or equal to 29 days after the study treatment administration
2-long terminal repeat (2LTR) circle DNA at baseline and after treatment | Measured through Week 48
Cell-associated HIV-1 RNA at baseline and after treatment | Measured through Week 48
RNA/DNA ratios in total CD4 cells at baseline and after treatment | Measured through Week 48
Expression of programmed cell death 1 ligand 2 (PD-L2) on dendritic cells and monocyte-derived macrophages | Measured through Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Eron Jr., MD, Study Chair — University of North Carolina, Chapel Hill
Locations (5):
- United States (5):
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Washington University Therapeutics (WT) CRS, St Louis, Missouri
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Cincinnati Clinical Research Site, Cincinnati, Ohio
  - Vanderbilt Therapeutics (VT) CRS, Nashville, Tennessee

REFERENCES:
- [Derived] Gay CL, Bosch RJ, Ritz J, Hataye JM, Aga E, Tressler RL, Mason SW, Hwang CK, Grasela DM, Ray N, Cyktor JC, Coffin JM, Acosta EP, Koup RA, Mellors JW, Eron JJ; AIDS Clinical Trials 5326 Study Team. Clinical Trial of the Anti-PD-L1 Antibody BMS-936559 in HIV-1 Infected Participants on Suppressive Antiretroviral Therapy. J Infect Dis. 2017 Jun 1;215(11):1725-1733. doi: 10.1093/infdis/jix191. PMID 28431010